CLINICAL TRIAL: NCT04867174
Title: COVID-19 Vaccination Take-Up in a County-Run Medicaid Managed Care Population
Brief Title: COVID-19 Vaccination Take-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: Contra Costa Health Services (Other Government); Abdul Latif Jameel Poverty Action Lab (Other); University of Southern California (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 27165; P30AG034532 (NIH)
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Covid19; Vaccination
Keywords: COVID19; vaccination
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Arm (Placebo Comparator): No messaging about COVID-19 vaccination
  Interventions: Behavioral: Financial incentives; Behavioral: Convenient scheduling link
- Emotional message (Experimental): Participants view an emotional video from the state of California about getting back to normal.
  Interventions: Behavioral: Financial incentives; Behavioral: Convenient scheduling link
- Safety and effectiveness message (Experimental): Participants view a video with information about the safety and effectiveness of the COVID-19 vaccines
  Interventions: Behavioral: Financial incentives; Behavioral: Convenient scheduling link; Behavioral: Race concordant; Behavioral: Gender concordant
- Consequences message (Experimental): Participants view a video with information about the consequences of not getting vaccinated against COVID-19.
  Interventions: Behavioral: Financial incentives; Behavioral: Convenient scheduling link; Behavioral: Race concordant; Behavioral: Gender concordant

INTERVENTIONS:
Behavioral: Financial incentives — Each of the study arms, including the no message/control arm, will be interacted with different financial incentives (N=5,000)
Behavioral: Convenient scheduling link — In addition, study arms will be randomly assigned a convenient link to the county public vaccine appointment scheduling system highlighted for participants (N=5,000).
Behavioral: Race concordant — Randomized to a messenger who is race concordant with the participant
  Arms: Consequences message; Safety and effectiveness message
Behavioral: Gender concordant — Randomized to a messenger who is gender concordant with the participant
  Arms: Consequences message; Safety and effectiveness message

SUMMARY:
In this work, the investigators are partnering with Contra Costa Health Services (CCHS), the department of health in Contra Costa County, CA, to measure COVID-19 vaccinations and other COVID-19 related preventive health behaviors in the county's Medicaid managed care population. This work will test ways to increase COVID-19 vaccine uptake. The investigators hypothesize that small financial incentives and other low-cost behavioral nudges can be used to increase vaccine uptake and reduce disparities in uptake among diverse racial/ethnic minority populations.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and over
* member of Contra Costa Health Plan (CCHP)

Exclusion Criteria:

* contraindications to vaccination, as determined by county health plan or other medical staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2701 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contra Costa Health Plan, Martinez, California, United States

IPD SHARING:
Plan to Share IPD: No
Our partner will not allow data sharing. Code will be shared.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a cross randomization design. Subjects were randomized equally to control (no message) or an emotional message, a safety/effectiveness message or a consequence message. Each message arm was further randomized to financial incentives [50%] vs. no financial incentives [50%], with 25% randomized to a $10 incentive and 25% to a $50 incentive Each arm further randomized to receive a convenient scheduling link highlighted [50%] vs. not [50%].
Groups:
- Safety Message; Discordant Gender and Race: Participants view a video with information about the safety and effectiveness of the COVID-19 vaccines. Race and gender of messenger were discordant with the participant.
- Consequences Message; Discordant Gender and Race: Participants view a video with information about the consequences of not getting vaccinated against COVID-19.
  Race and gender of messenger was discordant with the participant.
- Safety Message; Gender Concordant, Race Discordant: Participants view a video with information about the safety and effectiveness of the COVID-19 vaccines; gender concordant but race discordant messenger.
- Consequences Message; Gender Concordant, Race Discordant: Participants view a video with information about the consequences of not getting vaccinated against COVID-19; gender concordant but race discordant messenger.
- Safety Message; Gender Discordant and Race Concordant: Participants view a video with information about the safety and effectiveness of the COVID-19 vaccines; gender discordant but race concordant messenger.
- Consequences Message; Gender Discordant and Race Concordant: Participants view a video with information about the consequences of not getting vaccinated against COVID-19; gender discordant but race concordant messenger.
- Safety Message; Gender and Race Concordant: Participants view a video with information about the safety and effectiveness of the COVID-19 vaccines; gender and race concordant messenger.
- Consequences Message; Gender and Race Concordant: Participants view a video with information about the consequences of not getting vaccinated against COVID-19; gender and race concordant messenger.
- Link: Participants receive a link at the end of the survey to an easy vaccination scheduling system.
- Link and Emotional Message: Participants get a link and view the emotional message about getting back to normal.
- Link and Safety Message; Gender and Race Discordant: Participants receive a link to the easy vaccination scheduling system. Prior to this, participants view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender and race discordant messenger.
- Link and Consequences Message; Gender and Race Discordant: Participants receive a link to the easy vaccination scheduling system. Prior to this, participants view a video the consequences of not getting vaccinated against COVID-19 with a gender and race discordant messenger.
- Link; Safety Message; Gender Concordant and Race Discordant: Participants receive a link to the easy vaccination scheduling system. Prior to this, participants view a video the safety and effectiveness of the COVID-19 vaccines with a gender concordant and race discordant messenger.
- Link; Consequences Message; Gender Concordant and Race Discordant: Participants receive a link to the easy vaccination scheduling system. Prior to this, participants view a video the consequences of not getting vaccinated against COVID-19 with a gender concordant and race discordant messenger.
- Link; Safety Message; Gender Discordant and Race Concordant: Participants receive a link to the easy vaccination scheduling system. Prior to this, participants view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender discordant and race concordant messenger.
- Link; Consequences Message; Gender Discordant and Race Concordant: Participants receive a link to the easy vaccination scheduling system. Prior to this, participants view a video the consequences of not getting vaccinated against COVID-19 with a gender discordant and race concordant messenger.
- Link; Safety Message; Gender and Race Concordant: Participants receive a link to the easy vaccination scheduling system. Prior to this, participants view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender and race concordant messenger.
- Link and Consequences Message; Gender and Race Concordant: Participants receive a link to the easy vaccination scheduling system. Prior to this, participants view a video the consequences of not getting vaccinated against COVID-19 with a gender and race concordant messenger.
- $10 Financial Incentive: Participants offered a $10 financial incentive for vaccination.
- $10 Financial Incentive; Emotional Message: Participants offered a $10 financial incentive for getting vaccinated and view an emotional video from the state of California about getting back to normal.
- $10 Financial Incentive; Safety Message; Gender and Race Discordant: Participants offered a $10 financial incentive for vaccination and view a video with information about the safety and effectiveness of the COVID-19 vaccines; gender and race discordant messenger
- $10 Financial Incentive; Consequences Message; Gender and Race Discordant: Participants offered a $10 financial incentive and view a video with information about the consequences of not getting vaccinated against COVID-19; gender and race discordant messenger.
- $10 Financial Incentive; Safety Message; Gender Concordant and Race Discordant: Participants offered a $10 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines; gender concordant but race discordant messenger.
- $10 Financial Incentive; Consequences Message; Gender Concordant and Race Discordant: Participants offered a $10 financial incentive and view a video with information about the consequences of not getting vaccinated against COVID-19; gender concordant but race discordant messenger.
- $10 Financial Incentive; Safety Message; Gender Discordant and Race Concordant: Participants offered a $10 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines; gender discordant but race concordant messenger.
- $10 Financial Incentive; Consequences Message; Gender Discordant and Race Concordant: Participants offered a $10 financial incentive and view a video with information about the consequences of not getting vaccinated against COVID-19; gender discordant but race concordant messenger.
- $10 Financial Incentive; Safety Message; Gender and Race Concordant: Participants offered a $10 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines; gender and race concordant messenger.
- $10 Financial Incentive; Consequences Message; Gender and Race Concordant: Participants offered a $10 financial incentive and view a video with information about the consequences of not getting vaccinated against COVID-19 with a gender and race concordant messenger.
- $10 Financial Incentive; Link: Participants offered a $10 financial incentive and an easy vaccination scheduling link.
- $10 Financial Incentive; Link; Emotion Message: Participants offered a $10 financial incentive, a video message about getting back to normal, and an easy vaccination scheduling link.
- $10 Financial Incentive; Link; Safety Message, Gender and Race Discordant: Participants offered a $10 financial incentive, view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender and race discordant messenger and provided an easy vaccination scheduling link.
- $10 Financial Incentive; Link; Consequences Message, Gender and Race Discordant: Participants offered a $10 financial incentive, view a video with information about the consequences of not getting vaccination with a gender and race discordant messenger and provided an easy vaccination scheduling link.
- $10 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant: Participants offered a $10 financial incentive, view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender concordant and race discordant messenger and provided an easy vaccination scheduling link.
- $10 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant: Participants offered a $10 financial incentive, view a video with information about the consequences of not getting vaccinated with a gender concordant and race discordant messenger and provided an easy vaccination scheduling link.
- $10 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant: Participants offered a $10 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender discordant and race concordant messenger and provided an easy vaccination scheduling link.
- $10 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant: Participants offered a $10 financial incentive, view a video with information about the consequences of not getting vaccinated with a gender discordant and race concordant messenger and provided an easy vaccination scheduling link.
- $10 Financial Incentive; Link; Safety Message, Gender and Race Concordant: Participants offered a $10 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender and race concordant messenger and provided an easy vaccination scheduling link.
- $10 Financial Incentive; Link; Consequences Message, Gender and Race Concordant: Participants offered a $10 financial incentive and view a video with information about the consequences of not getting vaccinated against COVID-19 with a gender and race concordant messenger and provided an easy vaccination scheduling link
- $50 Financial Incentive: Participants offered a $50 financial incentive
- $50 Financial Incentive; Emotional Message: Participants offered a $50 financial incentive for getting vaccinated and view an emotional video from the state of California about getting back to normal.
- $50 Financial Incentive; Safety Message; Gender and Race Discordant: Participants offered a $10 financial incentive, view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender and race discordant messenger.
- $50 Financial Incentive; Consequences Message; Gender and Race Discordant: Participants offered a $50 financial incentive and view a video with information about the consequences of not getting vaccinated against COVID-19 with a gender and race discordant messenger.
- $50 Financial Incentive; Safety Message; Gender Concordant and Race Discordant: Participants offered a $50 financial incentive, view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender concordant and race discordant messenger.
- $50 Financial Incentive; Consequences Message; Gender Concordant and Race Discordant: Participants offered a $50 financial incentive for getting vaccinated and view a video with information about the consequences of not getting vaccinated against COVID-19 with a gender concordant and race discordant messenger.
- $50 Financial Incentive; Safety Message; Gender Discordant and Race Concordant: Participants offered a $50 financial incentive for getting vaccinated and view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender discordant and race concordant messenger.
- $50 Financial Incentive; Consequences Message; Gender Discordant and Race Concordant: Participants offered a $50 financial incentive for getting vaccinated and view a video with information about the consequences of not getting vaccinated against COVID-19 with a gender discordant and race concordant messenger.
- $50 Financial Incentive; Safety Message; Gender and Race Concordant: Participants offered a $50 financial incentive for getting vaccinated, view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender and race concordant messenger.
- $50 Financial Incentive; Consequences Message; Gender and Race Concordant: Participants offered a $50 financial incentive for getting vaccinated and view a video with information about the consequences of not getting vaccinated against COVID-19 with a gender and race concordant messenger.
- $50 Financial Incentive; Link: Participants offered a $50 financial incentive for getting vaccinated and provided an easy vaccination scheduling link.
- $50 Financial Incentive; Link; Emotion Message: Participants offered a $50 financial incentive for getting vaccinated, view an emotional video from the state of California about getting back to normal and provided an easy vaccination scheduling link.
- $50 Financial Incentive; Link; Safety Message, Gender and Race Discordant: Participants offered a $50 financial incentive for getting vaccinated, view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender and race discordant messenger and provided an easy vaccination scheduling link.
- $50 Financial Incentive; Link; Consequences Message, Gender and Race Discordant; $50 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant: Participants offered a $50 financial incentive for getting vaccinated, view a video with information about the consequences of not getting vaccinated against COVID-19 with a gender and race discordant messenger and provided an easy vaccination scheduling link.
- $50 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant: Participants offered a $50 financial incentive for getting vaccinated, view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender concordant and race discordant messenger and provided an easy vaccination scheduling link.
- $50 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant: Participants offered a $50 financial incentive for getting vaccinated, view a video with information about the consequences of not getting vaccinated against COVID-19 with a gender concordant and race discordant messenger and provided an easy vaccination scheduling link.
- $50 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant: Participants offered a $50 financial incentive for getting vaccinated, view a video with information about the safety and effectiveness of the COVID-19 vaccines with a discordant gender and race concordant messenger and provided an easy vaccination scheduling link.
- 50 Financial Incentive; Link; Safety Message, Gender and Race Concordant: Participants offered a $50 financial incentive for getting vaccinated, view a video with information about the safety and effectiveness of the COVID-19 vaccines with a gender and race concordant messenger and provided an easy vaccination scheduling link.
- 50 Financial Incentive; Link; Consequences Message, Gender and Race Concordant: Participants offered a $50 financial incentive for getting vaccinated and view a video with information about the consequences of not getting vaccinated against COVID-19 with a gender and race concordant messenger and provided an easy vaccination scheduling link.
Period: Overall Study
Arm/Group | Control Arm | Emotional Message | Safety Message; Discordant Gender and Race | Consequences Message; Discordant Gender and Race | Safety Message; Gender Concordant, Race Discordant | Consequences Message; Gender Concordant, Race Discordant | Safety Message; Gender Discordant and Race Concordant | Consequences Message; Gender Discordant and Race Concordant | Safety Message; Gender and Race Concordant | Consequences Message; Gender and Race Concordant | Link | Link and Emotional Message | Link and Safety Message; Gender and Race Discordant | Link and Consequences Message; Gender and Race Discordant | Link; Safety Message; Gender Concordant and Race Discordant | Link; Consequences Message; Gender Concordant and Race Discordant | Link; Safety Message; Gender Discordant and Race Concordant | Link; Consequences Message; Gender Discordant and Race Concordant | Link; Safety Message; Gender and Race Concordant | Link and Consequences Message; Gender and Race Concordant | $10 Financial Incentive | $10 Financial Incentive; Emotional Message | $10 Financial Incentive; Safety Message; Gender and Race Discordant | $10 Financial Incentive; Consequences Message; Gender and Race Discordant | $10 Financial Incentive; Safety Message; Gender Concordant and Race Discordant | $10 Financial Incentive; Consequences Message; Gender Concordant and Race Discordant | $10 Financial Incentive; Safety Message; Gender Discordant and Race Concordant | $10 Financial Incentive; Consequences Message; Gender Discordant and Race Concordant | $10 Financial Incentive; Safety Message; Gender and Race Concordant | $10 Financial Incentive; Consequences Message; Gender and Race Concordant | $10 Financial Incentive; Link | $10 Financial Incentive; Link; Emotion Message | $10 Financial Incentive; Link; Safety Message, Gender and Race Discordant | $10 Financial Incentive; Link; Consequences Message, Gender and Race Discordant | $10 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant | $10 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant | $10 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant | $10 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant | $10 Financial Incentive; Link; Safety Message, Gender and Race Concordant | $10 Financial Incentive; Link; Consequences Message, Gender and Race Concordant | $50 Financial Incentive | $50 Financial Incentive; Emotional Message | $50 Financial Incentive; Safety Message; Gender and Race Discordant | $50 Financial Incentive; Consequences Message; Gender and Race Discordant | $50 Financial Incentive; Safety Message; Gender Concordant and Race Discordant | $50 Financial Incentive; Consequences Message; Gender Concordant and Race Discordant | $50 Financial Incentive; Safety Message; Gender Discordant and Race Concordant | $50 Financial Incentive; Consequences Message; Gender Discordant and Race Concordant | $50 Financial Incentive; Safety Message; Gender and Race Concordant | $50 Financial Incentive; Consequences Message; Gender and Race Concordant | $50 Financial Incentive; Link | $50 Financial Incentive; Link; Emotion Message | $50 Financial Incentive; Link; Safety Message, Gender and Race Discordant | $50 Financial Incentive; Link; Consequences Message, Gender and Race Discordant | $50 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant | $50 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant | $50 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant | $50 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant | 50 Financial Incentive; Link; Safety Message, Gender and Race Concordant | 50 Financial Incentive; Link; Consequences Message, Gender and Race Concordant
Started | 136 | 137 | 29 | 37 | 32 | 31 | 43 | 33 | 39 | 35 | 147 | 122 | 30 | 31 | 30 | 23 | 35 | 34 | 34 | 27 | 113 | 103 | 27 | 22 | 30 | 24 | 33 | 28 | 17 | 32 | 117 | 100 | 20 | 19 | 28 | 15 | 22 | 22 | 24 | 18 | 112 | 120 | 28 | 18 | 26 | 33 | 21 | 20 | 21 | 23 | 104 | 99 | 28 | 23 | 27 | 26 | 19 | 30 | 20 | 24
Completed | 136 | 137 | 29 | 37 | 32 | 31 | 43 | 33 | 39 | 35 | 147 | 122 | 30 | 31 | 30 | 23 | 35 | 34 | 34 | 27 | 113 | 103 | 27 | 22 | 30 | 24 | 33 | 28 | 17 | 32 | 117 | 100 | 20 | 19 | 28 | 15 | 22 | 22 | 24 | 18 | 112 | 120 | 28 | 18 | 26 | 33 | 21 | 20 | 21 | 23 | 104 | 99 | 28 | 23 | 27 | 26 | 19 | 30 | 20 | 24
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a cross randomization design. Subjects were randomized equally to control (no message) or an emotional message, a safety/effectiveness message or a consequence message. Each of these arms was interacted with a financial incentive of $10 or $50 and, separately, with a convenient link to a vaccine appointment scheduling system. In practice, this means there are 60 arms. See protocol for details. Since it's not feasible to show all arms concisely, we report details by message arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Emotional Message | Safety Message; Discordant Gender and Race | Consequences Message; Discordant Gender and Race | Safety Message; Gender Concordant, Race Discordant | Consequences Message; Gender Concordant, Race Discordant | Safety Message; Gender Discordant and Race Concordant | Consequences Message; Gender Discordant and Race Concordant | Safety Message; Gender and Race Concordant | Consequences Message; Gender and Race Concordant | Link | Link and Emotional Message | Link and Safety Message; Gender and Race Discordant | Link and Consequences Message; Gender and Race Discordant | Link; Safety Message; Gender Concordant and Race Discordant | Link; Consequences Message; Gender Concordant and Race Discordant | Link; Safety Message; Gender Discordant and Race Concordant | Link; Consequences Message; Gender Discordant and Race Concordant | Link; Safety Message; Gender and Race Concordant | Link and Consequences Message; Gender and Race Concordant | $10 Financial Incentive | $10 Financial Incentive; Emotional Message | $10 Financial Incentive; Safety Message; Gender and Race Discordant | $10 Financial Incentive; Consequences Message; Gender and Race Discordant | $10 Financial Incentive; Safety Message; Gender Concordant and Race Discordant | $10 Financial Incentive; Consequences Message; Gender Concordant and Race Discordant | $10 Financial Incentive; Safety Message; Gender Discordant and Race Concordant | $10 Financial Incentive; Consequences Message; Gender Discordant and Race Concordant | $10 Financial Incentive; Safety Message; Gender and Race Concordant | $10 Financial Incentive; Consequences Message; Gender and Race Concordant | $10 Financial Incentive; Link | $10 Financial Incentive; Link; Emotion Message | $10 Financial Incentive; Link; Safety Message, Gender and Race Discordant | $10 Financial Incentive; Link; Consequences Message, Gender and Race Discordant | $10 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant | $10 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant | $10 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant | $10 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant | $10 Financial Incentive; Link; Safety Message, Gender and Race Concordant | $10 Financial Incentive; Link; Consequences Message, Gender and Race Concordant | $50 Financial Incentive | $50 Financial Incentive; Emotional Message | $50 Financial Incentive; Safety Message; Gender and Race Discordant | $50 Financial Incentive; Consequences Message; Gender and Race Discordant | $50 Financial Incentive; Safety Message; Gender Concordant and Race Discordant | $50 Financial Incentive; Consequences Message; Gender Concordant and Race Discordant | $50 Financial Incentive; Safety Message; Gender Discordant and Race Concordant | $50 Financial Incentive; Consequences Message; Gender Discordant and Race Concordant | $50 Financial Incentive; Safety Message; Gender and Race Concordant | $50 Financial Incentive; Consequences Message; Gender and Race Concordant | $50 Financial Incentive; Link | $50 Financial Incentive; Link; Emotion Message | $50 Financial Incentive; Link; Safety Message, Gender and Race Discordant | $50 Financial Incentive; Link; Consequences Message, Gender and Race Discordant | $50 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant | $50 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant | $50 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant | $50 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant | 50 Financial Incentive; Link; Safety Message, Gender and Race Concordant | 50 Financial Incentive; Link; Consequences Message, Gender and Race Concordant | Total
Number analyzed (Participants) | 136 | 137 | 29 | 37 | 32 | 31 | 43 | 33 | 39 | 35 | 147 | 122 | 30 | 31 | 30 | 23 | 35 | 34 | 34 | 27 | 113 | 103 | 27 | 22 | 30 | 24 | 33 | 28 | 17 | 32 | 117 | 100 | 20 | 19 | 28 | 15 | 22 | 22 | 24 | 18 | 112 | 120 | 28 | 18 | 26 | 33 | 21 | 20 | 21 | 23 | 104 | 99 | 28 | 23 | 27 | 26 | 19 | 30 | 20 | 24 | 2701
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.91 (11.73) | 34.82 (12.53) | 37.31 (14.70) | 39.32 (14.42) | 34.69 (10.20) | 36.65 (13.57) | 40.74 (14.39) | 40.30 (14.58) | 39.33 (14.80) | 37.46 (10.07) | 36.29 (12.03) | 38.37 (13.96) | 35.87 (13.05) | 34.03 (13.44) | 35.50 (9.31) | 37.39 (12.90) | 34.54 (13.54) | 34.15 (10.43) | 35.32 (10.31) | 39.11 (12.81) | 36.53 (12.51) | 33.83 (9.98) | 38.11 (17.34) | 34.14 (10.52) | 35.30 (12.80) | 36.79 (12.73) | 35.42 (12.75) | 35.14 (12.62) | 32.12 (13.26) | 37.97 (13.63) | 37.15 (12.92) | 33.99 (11.31) | 35.15 (16.52) | 29.63 (5.85) | 36.18 (11.10) | 32.80 (9.99) | 33.64 (12.03) | 34.77 (9.01) | 38.33 (14.61) | 39.67 (15.14) | 37.51 (12.28) | 36.87 (12.98) | 32.43 (10.02) | 39.78 (13.52) | 34.27 (11.53) | 40.64 (13.85) | 33.76 (11.10) | 37.45 (14.27) | 42.43 (16.74) | 34.35 (13.84) | 35.88 (11.63) | 37.93 (12.10) | 36.50 (10.73) | 33.70 (11.74) | 37.59 (14.13) | 38.12 (14.02) | 37.74 (14.96) | 35.50 (12.22) | 36.85 (12.49) | 37.63 (12.04) | 36.44 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 97 | 23 | 27 | 25 | 26 | 29 | 24 | 30 | 27 | 110 | 83 | 17 | 26 | 22 | 18 | 29 | 22 | 25 | 20 | 81 | 75 | 17 | 20 | 23 | 16 | 26 | 18 | 10 | 23 | 85 | 77 | 15 | 16 | 23 | 13 | 17 | 19 | 19 | 14 | 88 | 91 | 21 | 14 | 19 | 26 | 15 | 19 | 13 | 15 | 85 | 70 | 19 | 15 | 25 | 18 | 12 | 25 | 12 | 19 | 2007
  Male | 37 | 40 | 6 | 10 | 7 | 5 | 14 | 9 | 9 | 8 | 37 | 39 | 13 | 5 | 8 | 5 | 6 | 12 | 9 | 7 | 32 | 28 | 10 | 2 | 7 | 8 | 7 | 10 | 7 | 9 | 32 | 23 | 5 | 3 | 5 | 2 | 5 | 3 | 5 | 4 | 24 | 29 | 7 | 4 | 7 | 7 | 6 | 1 | 8 | 8 | 19 | 29 | 9 | 8 | 2 | 8 | 7 | 5 | 8 | 5 | 694
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (non-Hispanic) | 55 | 43 | 15 | 10 | 13 | 12 | 19 | 11 | 11 | 14 | 44 | 41 | 10 | 13 | 12 | 11 | 12 | 16 | 12 | 12 | 40 | 33 | 9 | 7 | 13 | 12 | 11 | 7 | 5 | 12 | 42 | 34 | 2 | 3 | 8 | 5 | 8 | 7 | 12 | 8 | 47 | 47 | 10 | 6 | 7 | 14 | 6 | 6 | 9 | 8 | 38 | 39 | 8 | 9 | 3 | 8 | 8 | 8 | 9 | 5 | 959
  Black (non-Hispanic) | 39 | 51 | 7 | 16 | 7 | 9 | 7 | 11 | 12 | 11 | 52 | 37 | 7 | 5 | 6 | 9 | 9 | 7 | 10 | 11 | 32 | 33 | 8 | 5 | 7 | 9 | 6 | 14 | 5 | 10 | 34 | 32 | 11 | 10 | 10 | 4 | 8 | 7 | 3 | 4 | 39 | 30 | 6 | 7 | 11 | 12 | 4 | 4 | 7 | 8 | 33 | 31 | 10 | 9 | 6 | 5 | 4 | 13 | 4 | 6 | 824
  Hispanic or Latino | 42 | 43 | 7 | 11 | 12 | 10 | 17 | 11 | 16 | 10 | 51 | 44 | 13 | 13 | 12 | 3 | 14 | 11 | 12 | 4 | 41 | 37 | 10 | 10 | 10 | 3 | 16 | 7 | 7 | 10 | 41 | 34 | 7 | 6 | 10 | 6 | 6 | 8 | 9 | 6 | 26 | 43 | 12 | 5 | 8 | 7 | 11 | 10 | 5 | 7 | 33 | 29 | 10 | 5 | 8 | 13 | 7 | 9 | 7 | 13 | 908

OUTCOME MEASURES:

1. Primary Outcome: Rate of COVID-19 Vaccination at 1 Month
Description: Percent of the population with at least one COVID-19 vaccination
Time Frame: 1 month
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Control Arm: Control, no videos, financial incentives or scheduling link.
- Safety Message; Discordant Gender and Race: Participants view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger has discordant Gender and Race.
- Consequences Message; Discordant Gender and Race: Participants view a video with information about the consequences of not getting vaccinated against COVID-19. Participant has discordant gender and race with messenger.
- Safety Message; Gender Concordant, Race Discordant: Participants view a video with info about safety and effectiveness of the vaccines. Messenger and Participant are Gender concordant but race discordant.
- Consequences Message; Gender Concordant and Race Discordant: Participants view a video with information about the consequences of not getting vaccinated against COVID-19. Participant has concordant gender but discordant race with messenger.
- Safety Message; Gender Discordant and Race Concordant: Participants view a video with info about safety and effectiveness of the vaccines. Messenger and Participant are Gender discordant but race concordant.
- Consequences Message; Gender Discordant and Race Concordant: Participants view a video with information about the consequences of not getting vaccinated against COVID-19. Participant has discordant gender but concordant race with messenger.
- Safety Message; Concordant Gender and Race: Participants view a video with info about safety and effectiveness of the vaccines. Messenger and Participant are Gender and race concordant.
- Consequences Message; Concordant Gender and Race: Participants view a video with information about the consequences of not getting vaccinated against COVID-19. Messenger and participant have concordant gender and race.
- Link: Participants receive a link at the end of the survey to an easy vaccine scheduling system.
- Link and Emotional Message: Participants receive an easy vaccine scheduling link and view an emotional video from the state of California about getting back to normal.
- Link and Safety Message; Gender and Race Discordant: Participants view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger has discordant Gender and Race. Receive link to easy vaccine scheduling tool.
- Link and Consequences Message; Gender and Race Discordant: Participants view a video about the consequences of not getting vaccinated. Messenger has discordant Gender and Race. Also receive link to an easy vaccine scheduling tool.
- Link and Safety Message; Gender Concordant and Race Discordant: Participants view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender concordant and Race discordant. Receive link to easy vaccine scheduling tool.
- Link and Consequences Message; Gender Concordant and Race Discordant: Participants view a video with information about the consequences of not getting vaccinated Messenger and Participant are Gender concordant and Race discordant. Receive link to easy vaccine scheduling tool.
- Link and Safety Message; Gender Discordant and Race Concordant: Participants view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender Discordant and Race Concordant. Receive link to easy vaccine scheduling tool.
- Link and Consequences Message; Gender Discordant and Race Concordant: Participants view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender Discordant and Race Concordant. Receive link to easy vaccine scheduling tool.
- Link and Safety Message; Gender and Race Concordant: Participants view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender and Race concordant. Receive link to easy vaccine scheduling tool.
- Link and Consequences Message; Gender and Race Concordant: Participants view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender and Race concordant. Receive link to easy vaccine scheduling tool.
- $10 Financial Incentive; Emotional Message: Participants offered $10 financial incentive for vaccination and view an emotional video from the state of California about getting back to normal.
- $10 Financial Incentive and Safety Message; Gender and Race Discordant: Participants offered a $10 incentive for vaccination and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender and Race discordant.
- $10 Financial Incentive and Consequences Message; Gender and Race Discordant: Participants offered a $10 vaccination incentive and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender and Race discordant.
- $10 Financial Incentive and Safety Message; Gender Concordant and Race Discordant: Participants offered a $10 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender Concordant and Race discordant.
- $10 Financial Incentive and Consequences Message; Gender Concordant and Race Discordant: Participants offered a $10 financial incentive and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender Concordant and Race discordant.
- $10 Financial Incentive and Safety Message; Gender Discordant and Race Concordant: Participants offered a $10 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender Discordant and Race Concordant.
- $10 Financial Incentive and Consequences Message; Gender Discordant and Race Concordant: Participants offered a $10 financial incentive and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender Discordant and Race Concordant.
- $10 Financial Incentive and Safety Message; Gender and Race Concordant: Participants offered a $10 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender and Race Concordant.
- $10 Financial Incentive and Consequences Message; Gender and Race Concordant: Participants offered a $10 financial incentive and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender and Race Concordant.
- $10 Financial Incentive; Link: Participant offered a $10 financial incentive for vaccination and given a link to an easy vaccination scheduling system.
- $10 Financial Incentive; Link; Emotional Message: Participants offered a $10 financial incentive for vaccination and view an emotional video from the state of California about getting back to normal.
- $10 Financial Incentive; Link; Safety Message; Gender and Race Discordant: Participants offered a $10 financial incentive for vaccination; receive link to easy vaccine scheduling tool and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender and Race discordant.
- $10 Financial Incentive; Link; Consequences Message, Gender and Race Discordant: Participants offered a $10 financial incentive for vaccination; receive link to easy vaccine scheduling tool and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender and Race discordant.
- $10 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant: Participants offered a $10 financial incentive, given a link to an easy vaccination scheduling system and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender Concordant and Race Discordant.
- $10 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant: Participants offered a $10 financial incentive for vaccination; receive link to easy vaccine scheduling tool and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender Concordant and Race discordant.
- $10 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant; $10 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant: Participants offered a $10 financial incentive for vaccination; receive link to easy vaccine scheduling tool and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender Discordant and Race Concordant.
- $10 Financial Incentive; Link; Safety Message, Gender and Race Concordant; $10 Financial Incentive; Link; Consequences Message, Gender and Race Concordant: Participants offered a $10 financial incentive for vaccination; receive link to easy vaccine scheduling tool and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender and Race Concordant.
- $50 Financial Incentive: Participants offered a $50 financial incentive for vaccination.
- $50 Financial Incentive; Emotional Message: Participants offered a $50 financial incentive for vaccination; view an emotional video from the state of California about getting back to normal.
- $50 Financial Incentive; Safety Message; Gender and Race Discordant: Participants offered a $50 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender and Race discordant.
- $50 Financial Incentive; Consequences Message; Gender and Race Discordant: Participants offered a $50 financial incentive and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender and Race discordant.
- $50 Financial Incentive; Safety Message; Gender Concordant and Race Discordant: Participants offered a $50 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender Concordant and Race discordant.
- $50 Financial Incentive; Consequences Message; Gender Concordant and Race Discordant: Participants offered a $50 financial incentive and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender Concordant and Race discordant.
- $50 Financial Incentive; Safety Message; Gender Discordant and Race Concordant: Participants offered a $50 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender discordant and Race concordant.
- $50 Financial Incentive; Consequences Message; Gender Discordant and Race Concordant: Participants offered a $50 financial incentive and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender discordant and Race concordant.
- $50 Financial Incentive; Safety Message; Gender and Race Concordant: Participants offered a $50 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender and Race concordant.
- $50 Financial Incentive; Consequences Message; Gender and Race Concordant: Participants offered a $50 financial incentive and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender and Race Concordant.
- $50 Financial Incentive; Link: Participant offered a $50 financial incentive for vaccination and given a link to an easy vaccination scheduling system.
- $50 Financial Incentive; Link; Emotional Message: Participants offered $50 financial incentive for vaccination; receive an easy vaccine scheduling link and view an emotional video from the state of California about getting back to normal.
- $50 Financial Incentive; Link; Safety Message, Gender and Race Discordant: Participants offered a $50 financial incentive and view a video with information about the safety and effectiveness of the COVID-19 vaccines. They receive a link to an easy vaccination scheduling system. Messenger and Participant are Gender and Race discordant.
- $50 Financial Incentive; Link; Consequences Message, Gender and Race Discordant: Participants offered a $50 financial incentive and given a link to an easy vaccine scheduling system. Participants view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender and Race discordant.
- $50 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant: Participant offered a $50 financial incentive for vaccination and given a link to an easy vaccination scheduling system. They view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender Concordant and Race discordant.
- $50 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant: Participants offered a $50 financial incentive for vaccination; receive link to easy vaccine scheduling tool and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender concordant and Race discordant.
- $50 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant: Participants offered a $50 financial incentive, given a link to an easy vaccination scheduling system and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender discordant and Race concordant.
- $50 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant: Participants offered a $50 financial incentive for vaccination; receive link to easy vaccine scheduling tool and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender discordant and Race concordant.
- 50 Financial Incentive; Link; Safety Message, Gender and Race Concordant: Participants offered a $50 financial incentive, given a link to an easy vaccination scheduling system and view a video with information about the safety and effectiveness of the COVID-19 vaccines. Messenger and Participant are Gender and Race concordant.
- 50 Financial Incentive; Link; Consequences Message, Gender and Race Concordant: Participants offered a $50 financial incentive for vaccination; receive link to easy vaccine scheduling tool and view a video with information about the consequences of not getting vaccinated. Messenger and Participant are Gender and Race concordant.
Arm/Group | Control Arm | Emotional Message | Safety Message; Discordant Gender and Race | Consequences Message; Discordant Gender and Race | Safety Message; Gender Concordant, Race Discordant | Consequences Message; Gender Concordant and Race Discordant | Safety Message; Gender Discordant and Race Concordant | Consequences Message; Gender Discordant and Race Concordant | Safety Message; Concordant Gender and Race | Consequences Message; Concordant Gender and Race | Link | Link and Emotional Message | Link and Safety Message; Gender and Race Discordant | Link and Consequences Message; Gender and Race Discordant | Link and Safety Message; Gender Concordant and Race Discordant | Link and Consequences Message; Gender Concordant and Race Discordant | Link and Safety Message; Gender Discordant and Race Concordant | Link and Consequences Message; Gender Discordant and Race Concordant | Link and Safety Message; Gender and Race Concordant | Link and Consequences Message; Gender and Race Concordant | $10 Financial Incentive | $10 Financial Incentive; Emotional Message | $10 Financial Incentive and Safety Message; Gender and Race Discordant | $10 Financial Incentive and Consequences Message; Gender and Race Discordant | $10 Financial Incentive and Safety Message; Gender Concordant and Race Discordant | $10 Financial Incentive and Consequences Message; Gender Concordant and Race Discordant | $10 Financial Incentive and Safety Message; Gender Discordant and Race Concordant | $10 Financial Incentive and Consequences Message; Gender Discordant and Race Concordant | $10 Financial Incentive and Safety Message; Gender and Race Concordant | $10 Financial Incentive and Consequences Message; Gender and Race Concordant | $10 Financial Incentive; Link | $10 Financial Incentive; Link; Emotional Message | $10 Financial Incentive; Link; Safety Message; Gender and Race Discordant | $10 Financial Incentive; Link; Consequences Message, Gender and Race Discordant | $10 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant | $10 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant | $10 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant | $10 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant | $10 Financial Incentive; Link; Safety Message, Gender and Race Concordant | $10 Financial Incentive; Link; Consequences Message, Gender and Race Concordant | $50 Financial Incentive | $50 Financial Incentive; Emotional Message | $50 Financial Incentive; Safety Message; Gender and Race Discordant | $50 Financial Incentive; Consequences Message; Gender and Race Discordant | $50 Financial Incentive; Safety Message; Gender Concordant and Race Discordant | $50 Financial Incentive; Consequences Message; Gender Concordant and Race Discordant | $50 Financial Incentive; Safety Message; Gender Discordant and Race Concordant | $50 Financial Incentive; Consequences Message; Gender Discordant and Race Concordant | $50 Financial Incentive; Safety Message; Gender and Race Concordant | $50 Financial Incentive; Consequences Message; Gender and Race Concordant | $50 Financial Incentive; Link | $50 Financial Incentive; Link; Emotional Message | $50 Financial Incentive; Link; Safety Message, Gender and Race Discordant | $50 Financial Incentive; Link; Consequences Message, Gender and Race Discordant | $50 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant | $50 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant | $50 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant | $50 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant | 50 Financial Incentive; Link; Safety Message, Gender and Race Concordant | 50 Financial Incentive; Link; Consequences Message, Gender and Race Concordant
Number analyzed (Participants) | 136 | 137 | 29 | 37 | 32 | 31 | 43 | 33 | 39 | 35 | 147 | 122 | 30 | 31 | 30 | 23 | 35 | 34 | 34 | 27 | 113 | 103 | 27 | 22 | 30 | 24 | 33 | 28 | 17 | 32 | 117 | 100 | 20 | 19 | 28 | 15 | 22 | 22 | 24 | 18 | 112 | 120 | 28 | 18 | 26 | 33 | 21 | 20 | 21 | 23 | 104 | 99 | 28 | 23 | 27 | 26 | 19 | 30 | 20 | 24
Participants
  Number of Particpants who Received Vaccine | 12 | 4 | 0 | 1 | 2 | 3 | 3 | 3 | 3 | 3 | 15 | 17 | 2 | 1 | 3 | 2 | 2 | 2 | 4 | 1 | 10 | 5 | 3 | 2 | 3 | 1 | 3 | 0 | 1 | 3 | 9 | 6 | 0 | 1 | 2 | 1 | 0 | 1 | 3 | 1 | 6 | 13 | 9 | 1 | 3 | 4 | 1 | 0 | 1 | 1 | 4 | 9 | 2 | 1 | 0 | 4 | 0 | 1 | 2 | 2
  Number of Participants who did not Receive Vaccine | 124 | 133 | 29 | 36 | 30 | 28 | 40 | 30 | 36 | 32 | 132 | 105 | 28 | 30 | 27 | 21 | 33 | 32 | 30 | 26 | 103 | 98 | 24 | 20 | 27 | 23 | 30 | 28 | 16 | 29 | 108 | 94 | 20 | 18 | 26 | 14 | 22 | 21 | 21 | 17 | 106 | 107 | 19 | 17 | 23 | 29 | 20 | 20 | 20 | 22 | 100 | 90 | 26 | 22 | 27 | 22 | 19 | 29 | 18 | 22

2. Other Pre Specified Outcome: Vaccine Intentions
Description: Stated intention of receiving COVID-19 vaccination in the next 30 days (0% - 100% probability)
Time Frame: 30 days
Population: This is a cross randomization design. Subjects were randomized equally to control (no message) or an emotional message, a safety/effectiveness message or a consequence message. Each ofthese arms was interacted with a fi nancial incentive of $10 or $50 and, separately, with a convenient link to a vaccine appointment scheduling system. In practice, this means there are 60 arms.See protocol for details
Measure: Mean (Standard Deviation); unit: percent probability
Arm/Group | Control Arm | Emotional Message | Safety Message; Discordant Gender and Race | Consequences Message; Discordant Gender and Race | Safety Message; Gender Concordant, Race Discordant | Consequences Message; Gender Concordant and Race Discordant | Safety Message; Gender Discordant and Race Concordant | Consequences Message; Gender Discordant and Race Concordant | Safety Message; Concordant Gender and Race | Consequences Message; Concordant Gender and Race | Link | Link and Emotional Message | Link and Safety Message; Gender and Race Discordant | Link and Consequences Message; Gender and Race Discordant | Link and Safety Message; Gender Concordant and Race Discordant | Link and Consequences Message; Gender Concordant and Race Discordant | Link and Safety Message; Gender Discordant and Race Concordant | Link and Consequences Message; Gender Discordant and Race Concordant | Link and Safety Message; Gender and Race Concordant | Link and Consequences Message; Gender and Race Concordant | $10 Financial Incentive | $10 Financial Incentive; Emotional Message | $10 Financial Incentive and Safety Message; Gender and Race Discordant | $10 Financial Incentive and Consequences Message; Gender and Race Discordant | $10 Financial Incentive and Safety Message; Gender Concordant and Race Discordant | $10 Financial Incentive and Consequences Message; Gender Concordant and Race Discordant | $10 Financial Incentive and Safety Message; Gender Discordant and Race Concordant | $10 Financial Incentive and Consequences Message; Gender Discordant and Race Concordant | $10 Financial Incentive and Safety Message; Gender and Race Concordant | $10 Financial Incentive and Consequences Message; Gender and Race Concordant | $10 Financial Incentive; Link | $10 Financial Incentive; Link; Emotional Message | $10 Financial Incentive; Link; Safety Message; Gender and Race Discordant | $10 Financial Incentive; Link; Consequences Message, Gender and Race Discordant | $10 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant | $10 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant | $10 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant | $10 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant | $10 Financial Incentive; Link; Safety Message, Gender and Race Concordant | $10 Financial Incentive; Link; Consequences Message, Gender and Race Concordant | $50 Financial Incentive | $50 Financial Incentive; Emotional Message | $50 Financial Incentive; Safety Message; Gender and Race Discordant | $50 Financial Incentive; Consequences Message; Gender and Race Discordant | $50 Financial Incentive; Safety Message; Gender Concordant and Race Discordant | $50 Financial Incentive; Consequences Message; Gender Concordant and Race Discordant | $50 Financial Incentive; Safety Message; Gender Discordant and Race Concordant | $50 Financial Incentive; Consequences Message; Gender Discordant and Race Concordant | $50 Financial Incentive; Safety Message; Gender and Race Concordant | $50 Financial Incentive; Consequences Message; Gender and Race Concordant | $50 Financial Incentive; Link | $50 Financial Incentive; Link; Emotional Message | $50 Financial Incentive; Link; Safety Message, Gender and Race Discordant | $50 Financial Incentive; Link; Consequences Message, Gender and Race Discordant | $50 Financial Incentive; Link; Safety Message, Gender Concordant and Race Discordant | $50 Financial Incentive; Link; Consequences Message, Gender Concordant and Race Discordant | $50 Financial Incentive; Link; Safety Message, Gender Discordant and Race Concordant | $50 Financial Incentive; Link; Consequences Message, Gender Discordant and Race Concordant | 50 Financial Incentive; Link; Safety Message, Gender and Race Concordant | 50 Financial Incentive; Link; Consequences Message, Gender and Race Concordant
Number analyzed (Participants) | 136 | 137 | 29 | 37 | 32 | 31 | 43 | 33 | 39 | 35 | 147 | 122 | 30 | 31 | 30 | 23 | 35 | 34 | 34 | 27 | 113 | 103 | 27 | 22 | 30 | 24 | 33 | 28 | 17 | 32 | 117 | 100 | 20 | 19 | 28 | 15 | 22 | 22 | 24 | 18 | 112 | 120 | 28 | 18 | 26 | 33 | 21 | 20 | 21 | 23 | 104 | 99 | 28 | 23 | 27 | 26 | 19 | 30 | 20 | 24
percent probability | 34.13 (33.80) | 37.87 (33.85) | 29.31 (31.79) | 46.11 (30.13) | 38.72 (32.19) | 41.61 (30.53) | 40.60 (36.28) | 35.24 (33.88) | 37.36 (37.55) | 48.49 (34.50) | 37.88 (33.48) | 39.34 (31.67) | 42.30 (33.92) | 39.77 (31.81) | 46.07 (30.16) | 40.96 (36.18) | 37.89 (33.10) | 38.76 (38.81) | 31.91 (34.83) | 39.07 (37.83) | 33.02 (31.83) | 34.76 (33.39) | 36.26 (33.22) | 40.86 (28.73) | 49.17 (37.82) | 46.17 (36.27) | 41.24 (31.30) | 42.96 (29.47) | 44.29 (32.14) | 47.63 (31.79) | 35.72 (32.84) | 41.67 (34.33) | 30.25 (26.25) | 32.26 (36.41) | 42.79 (40.32) | 34.87 (24.36) | 35.36 (32.74) | 41.68 (36.42) | 42.29 (38.97) | 45.28 (39.08) | 29.67 (29.39) | 36.12 (32.55) | 48.07 (38.34) | 36.33 (35.22) | 33.38 (28.73) | 50.64 (36.10) | 37.24 (22.78) | 58.15 (31.55) | 42.76 (36.24) | 48.13 (33.91) | 32.32 (31.79) | 33.26 (31.11) | 45.86 (37.32) | 50.70 (30.45) | 31.22 (30.38) | 39.31 (36.02) | 41.11 (35.37) | 38.33 (30.85) | 45.40 (34.78) | 35.75 (30.03)

ADVERSE EVENTS:
Time Frame: 1 month from survey completion
Description: No difference. Cross randomization design. Subjects were randomized equally to control (no message) or an emotional message, a safety/effectiveness message or a consequence message. Each of these arms was interacted with a financial incentive of $10 or $50 and, separately, with a convenient link to a vaccine appointment scheduling system. In practice, this means there are 60 arms. See protocol for details. Since it's not feasible to show all arms concisely, we report details by message arm.
Groups:
- Control Arm: No messaging about COVID-19 vaccination
  Financial incentives: Interaction with $10 and $50 financial incentives.
  Convenient scheduling link: Interaction with a convenient link to the county public vaccine appointment scheduling system.
- Emotional Message: Participants view an emotional video from the state of California about getting back to normal.
  Financial incentives: Interaction with $10 and $50 financial incentives.
  Convenient scheduling link: Interaction with a convenient link to the county public vaccine appointment scheduling system.
- Safety and Effectiveness Message: Participants view a video with information about the safety and effectiveness of the COVID-19 vaccines
  Financial incentives: Interaction with $10 and $50 financial incentives.
  Convenient scheduling link: Interaction with a convenient link to the county public vaccine appointment scheduling system.
- Consequences Message: Participants view a video with information about the consequences of not getting vaccinated against COVID-19.
  Financial incentives: Interaction with $10 and $50 financial incentives.
  Convenient scheduling link: Interaction with a convenient link to the county public vaccine appointment scheduling system.
Arm/Group | Control Arm | Emotional Message | Safety and Effectiveness Message | Consequences Message
All-Cause Mortality (participants affected / at risk) | 0/729 | 0/681 | 0/663 | 0/628
Serious Adverse Events (participants affected / at risk) | 0/729 | 0/681 | 0/663 | 0/628
Other Adverse Events (participants affected / at risk) | 0/729 | 0/681 | 0/663 | 0/628

LIMITATIONS AND CAVEATS:
Enrollment was lower than initial anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT04867174/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT04867174/SAP_000.pdf